CLINICAL TRIAL: NCT01920360
Title: Study of the Effects of Immersion Baths in Sulphurous Water in Patients With Knee Osteoarthritis: Randomized Controlled Clinical Trial.
Brief Title: Evaluation Study of the Effects of Sulphurous Water in the Treatment of Knee Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Marcelo Branco, physiotherapist, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 65463
Record Dates: First submitted 2013-08-01; First posted 2013-08-12 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: KNEE OSTEOARTHRITIS
Keywords: KNEE OSTEOARTHRITIS; BALNEOTHERAPY; SULPHUROUS WATERS; WOMAC; LEQUESNE; HEALTH ASSESSMENT QUESTIONNAIRE; SHORT FORM - 36; VAS
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Balneology; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SULPHUROUS WATERS IMMERSION BATHS (Experimental): The baths will be held in individual tubs, properly disinfected, supplied with sulphurous thermal water at a temperature 37-39 ° C, which encompass the optimum temperatures for therapeutic bath. The baths lasted for 20 minutes. The subjects will drink two cups of water, 300 ml before and after the baths, in order to avoid an imbalance water.
  Interventions: Other: SULPHUROUS WATERS IMMERSION BATHS
- NOT SULPHUROUS WATERS IMMERSION BATHS (Experimental): The baths will be held in individual tubs, properly disinfected, supplied with not sulphurous thermal water at a temperature 37-39 ° C, which encompass the optimum temperatures for therapeutic bath. The baths lasted for 20 minutes. The subjects will drink two cups of water, 300 ml before and after the baths, in order to avoid an imbalance water.
  Interventions: Other: NOT SULPHUROUS WATERS IMMERSION BATHS
- CONTROL GROUP (Experimental): This group did not receive any treatment, only received some verbal directions as to the care that should be taken to prevent and control the knee pain.
  Interventions: Other: CONTROL GROUP

INTERVENTIONS:
Other: SULPHUROUS WATERS IMMERSION BATHS — SULPHUROUS WATERS IMMERSION BATHS: The baths will be held in individual tubs, properly disinfected, supplied with sulphurous thermal water at a temperature 37-39 ° C, which encompass the optimum temperatures for therapeutic bath. The baths lasted for 20 minutes. The subjects will drink two cups of water, 300 ml before and after the baths, in order to avoid an imbalance water.
  Other Names: Balneotherapy; Termalism
  Arms: SULPHUROUS WATERS IMMERSION BATHS
Other: NOT SULPHUROUS WATERS IMMERSION BATHS — NOT SULPHUROUS WATERS IMMERSION BATHS:The baths will be held in individual tubs, properly disinfected, supplied with not sulphur thermal water at a temperature 37-39 ° C, which encompass the optimum temperatures for therapeutic bath. The baths lasted for 20 minutes. The subjects will drink two cups of water, 300 ml before and after the baths, in order to avoid an imbalance water.
  Other Names: Balneotherapy; Termalism
  Arms: NOT SULPHUROUS WATERS IMMERSION BATHS
Other: CONTROL GROUP — CONTROL GROUP: This group did not receive any treatment, only received some verbal directions as to the care that should be taken to prevent and control the knee pain.
  Arms: CONTROL GROUP

SUMMARY:
The objectives are to evaluate the effects of immersion bath with sulphurous water in pain, joint mobility and quality of life in patients with knee osteoarthritis. Patients will undergo three weekly baths in sulphurous water and not sulphurous, twenty minutes each, for ten weeks.

The expected results are: reduction of pain, improved range of motion of the lower limbs with consequent increase in muscle mass improvement in postural balance, which will come due to the reduction of pain and improvement movements of the lower limbs; greater independence in performing the activities of daily living, better quality of life.

DETAILED DESCRIPTION:
The baths were performed in individual tubs, properly disinfected, supplied with thermal water and sulphurous thermal sulphurous not at a temperature 37-39 ° C, which encompass the optimum temperatures for therapeutic bath. The baths lasted for 20 minutes. The subjects drank two cups of water, 300 ml before and after the baths, in order to avoid an imbalance water. Treatment consisted of 30 individual treatment sessions, three times a week, lasting twenty minutes each session, for ten weeks. The experiment was performed at the Therms Antonio Carlos, institution belonging to the Municipality of Poços de Caldas, Minas Gerais, Brazil.

ELIGIBILITY:
Inclusion Criteria:

We selected individuals of both genders, diagnosed with Osteoarthritis of the knee according to the classification criteria of the American College of Rheumatology (ACR) only grades I to III chronic pain at some knees, for a minimum period of three months.

Exclusion Criteria:

* Patients with fibromyalgia;
* Individuals with respiratory diseases;
* Rheumatic diseases autoimmune inflammatory;
* Patients with uncontrolled thyroidopathies;
* Patients with injuries or amputations of lower limbs;
* Patients with psychiatric disorders or cognitive;
* Patients with a history of osteoporotic fracture;
* Patients with malignant
* Patients with infectious processes;
* Patients pregnant;
* Individuals who failed to enter the baths due to physical limitations;
* Were also excluded those who were engaged in other forms of treatment or using painkillers and anti-inflammatory drugs for other diseases. Note: were not excluded participants who were diagnosed with osteoarthritis in the spine, herniated, or degenerative disc protrusions.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-02; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pain | 10 weeks
  Tools:
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC): 5 questions about pain, 2 about stiffness, 17 about physical function. Each question receives a score from 0 to 100. After is done the arithmetic mean. The higher the score on each subscale, the greater deficit.
  Visual Analogic Scale (VAS): horizontal line marked from 0 (no pain) to 10 (intense pain).
  LEQUESNE: 11 questions about pain, discomfort and function, 6 about pain and discomfort, 1 about to walk away, and 4 on daily activities. The scores range from 0 (no impairment) to 24 (severe).
  Short Form-36 (SF-36): 36 items grouped into eight areas. The final score from 0 (worst quality) to 100 (the best).
Life Quality | 10 weeks
  Tools:
  Short Form-36 (SF-36): 36 items grouped into eight areas. The final score from 0 (worst quality) to 100 (the best).
Physical Function | 10 weeks
  Tools:
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC): 5 questions about pain, 2 about stiffness, 17 about physical function. Each question receives a score from 0 to 100. After is done the arithmetic mean. The higher the score on each subscale, the greater deficit.
  LEQUESNE: 11 questions about pain, discomfort and function, 6 about pain and discomfort, 1 about to walk away, and 4 on daily activities. The scores range from 0 (no impairment) to 24 (severe).
  Health Assessment Questionnaire (HAQ): Each question ranges from zero (no functional impairment) to three (task disabling).
  Short Form-36 (SF-36): 36 items grouped into eight areas. The final score from 0 (worst quality) to 100 (the best).

SECONDARY OUTCOMES:
Intake of pain medication | 10 weeks
  After randomization, patients were instructed to report home about taking medication for pain in the knees, noting in a spreadsheet every time you wear some medicine to relieve pain in the knees. The result of this analysis was based on the number of times each individual ingested some medication.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Branco, Principal Investigator — Federal University of São Paulo UNIFESP
Locations (1):
- Therms Antonio Carlos, Poços de Caldas, Minas Gerais, Brazil

REFERENCES:
- [Background] Verhagen AP, Bierma-Zeinstra SM, Boers M, Cardoso JR, Lambeck J, de Bie RA, de Vet HC. Balneotherapy for osteoarthritis. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD006864. doi: 10.1002/14651858.CD006864. PMID 17943920
- [Result] Yurtkuran M, Yurtkuran M, Alp A, Nasircilar A, Bingol U, Altan L, Sarpdere G. Balneotherapy and tap water therapy in the treatment of knee osteoarthritis. Rheumatol Int. 2006 Nov;27(1):19-27. doi: 10.1007/s00296-006-0158-8. Epub 2006 Jul 11. PMID 16832639